CLINICAL TRIAL: NCT04441632
Title: The Impact of Positive Reinforcement on Teamwork Climate, Resiliency, and Burnout During the COVID-19 Pandemic: the TEAM-ICU Study (Transforming Employee Attitudes Via Messaging Strengthens Interconnection, Communication, and Unity)
Brief Title: Effect of Positive Attitudes on Behavior and Wellness
Acronym: TEAM-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jack Green, Assistant Professor of Pediatrics, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000786
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Burnout; Stress, Emotional
Keywords: wellness; healthcare; burnout; COVID
MeSH Terms: conditions — Burnout, Psychological; Stress, Psychological | interventions — Feedback, Physiological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive feedback (Other): Participants in the study will provide consistent positive feedback to the colleagues they work with in the medical ICU (MICU) over a 4 week duration.
  Interventions: Behavioral: Positive feedback

INTERVENTIONS:
Behavioral: Positive feedback — Participants will submit positive feedback comments to their colleagues (anonymously or signed, participant-dependent) through an anonymous survey link, a minimum of twice weekly to 6 uniquely different individuals over a 4 week period (total minimum 24 unique individuals over the study period).

SUMMARY:
The COVID-19 pandemic has undoubtedly elevated levels of stress to people all over the globe, but none more than to the providers on the front-line. The purpose of the study is to first, assess the effects of the pandemic on burnout, team cohesion, and resiliency among healthcare providers battling COVID-19 together in a medical ICU (MICU). Secondly, the investigators hope to then assess the effects of simple positive feedback on transforming culture and attitudes during times of major stress.

ELIGIBILITY:
Inclusion Criteria:

* Front-line healthcare providers in the Medical Intensive Care Unit (MICU): nurses, respiratory therapists, resident physicians, fellow physicians, and attending physicians

Exclusion Criteria:

* Healthcare providers providing only consultatory care in the MICU
* Front-line healthcare providers not working in the MICU during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Teamwork climate, as measured by selected items from the validated Safety Attitude Questionnaire (SAQ) | 4 weeks
  The SAQ measures teamwork climate, safety climate, job satisfaction, stress recognition, perceptions of management, and working conditions. The six items assessing teamwork climate will be used. 5 point likert scale is used. Mean of the items - 1 * 25 will convert each participant's results to a 100 point scale (0, 25, 50, 75, 100 points).
Resiliency, as measured by the validated Brief Resilience Scale (BRS) | 4 weeks
  The BRS is comprised of 6 items on a likert scale. Responses varying from 1-5 for all six items give a total range of 6-30. This sum will be divided by the total number of questions for a final score.
Burnout, as validated by the single-item burnout scale inventory | 4 weeks
  This single item inventory provides 5 definitions of burnout that the participant will choose that most closely fits their personal level of burnout at the moment

CONTACTS AND LOCATIONS:
Overall Officials: Jack Green, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No